CLINICAL TRIAL: NCT05492929
Title: The Effect of Deep Breathing Exercise and 4-7-8 Breathing Techniques Applied to Patients After Bariatric Surgery on Anxiety and Quality of Life
Brief Title: The Effect of Deep Breathing Exercise and 4-7-8 Breathing Techniques on Anxiety and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Vesile Eskici Ilgin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: vesile18
Record Dates: First submitted 2022-08-04; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Complications
Keywords: 4-7-8 breathing technique; anxiety; bariatric surgery; deep breathing exercise; quality of life
MeSH Terms: conditions — Postoperative Complications; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The deep breathing group (Experimental): The deep breathing group was administered the nightly state and trait anxiety scale and SAAQ before the operation, and then they were informed about the deep breathing exercise. Between the 1st and 6th hours of the postoperative period, deep breathing exercise was performed, with 10 breaths per hour. At the end of the 6th hour, the state anxiety scale and SSWS were administered.
  Interventions: Other: The deep breathing group
- 4-7-8 breathing technique Group (Experimental): The nightly state and trait anxiety scale and the PSSQ were applied to the 4-7-8 breathing group before the operation, and then they were given information about the 4-7-8 breathing technique. Between the 1st and 6th hours postoperatively, the 4-7-8 breathing technique was applied for 1 set (4 breaths) every hour. At the end of the 6th hour, the state anxiety scale and SSWS were administered.
  Interventions: Other: 4-7-8 breathing technique
- control group (No Intervention): In the control group, the nightly state and trait anxiety scale and PSSQ were applied before the operation. At the end of the 6th hour postoperatively, without any application, the state anxiety scale and PSSQ were applied.

INTERVENTIONS:
Other: The deep breathing group — The deep breathing group
  Arms: The deep breathing group
Other: 4-7-8 breathing technique — 4-7-8 breathing technique Group
  Arms: 4-7-8 breathing technique Group

SUMMARY:
Aim: This study aims to determine the effects of the deep breathing exercise and the 4-7-8 breathing technique applied to patients after bariatric surgery on their anxiety and quality of life.

Materials and Methods: The study was conducted between January and June 2022 at Ankara Lokman Hekim Akay Hospital Endocrinology and Metabolic Diseases Clinic. The research was carried out using the pre-test post-test randomized controlled experimental research design with a control group. A total of 90 patients (30 patients in the deep breathing group, 30 patients in the 4-7-8 breathing group, and 30 patients in the control group) who met the research inclusion criteria were included in the study. While routine care was applied to the control group, 1 group was given deep breathing training, and the other group was given 4-7-8 breathing training. Personal Information Form, the Obesity-Specific Quality of Life Questionnaire, Status, and the State-Trait Anxiety Inventory were used for data collection. In the evaluation of the data, number, percentage, mean, standard deviation, Kolmogorov Smirnov test, chi- square, dependent samples t-test, ANOVA, Tukey's test, Pearson Correlation analysis, and Cronbach's alpha Reliability Coefficient were used.

DETAILED DESCRIPTION:
Obesity is a disease whose prevalence is increasing all over the world, reducing the quality and duration of life. Obesity affects the quality of life in all areas, including physiological, psychological, social and environmental aspects. Obesity causes anxiety, depression, low self-esteem and low body image in individuals. Obesity Bariatric surgery is considered to be the most effective and permanent method for weight loss in the treatment of cancer.

In the first month after bariatric surgery, unexpected conditions such as bleeding, thromboembolism, anastomotic leakage, and atelectasis may develop. In obese individuals, lung compliance decreases due to increased pulmonary blood volume and collapse in the peripheral airways. At the same time, excess adipose tissue accumulated in the chest wall and abdomen compresses the thorax and diaphragm, reducing lung volume. Positioning to relieve breathing, in-bed rotation movements, deep breathing and coughing exercises are the most important parts of nursing care, and interventions to prevent pulmonary complications in the postoperative period.

Anxiety is the whole of the natural reactions developed by the body and mind in the face of a situation or stimulus that disturbs the individual and endanger the existence. In everyday language, anxiety is expressed as anxiety and distress.

Gariepy et al. In a review by, it was seen that there is a positive relationship between obesity and anxiety disorders in general. Studies have shown that patients who are suitable for bariatric surgery among obese individuals have high levels of anxiety and depression, and generally have psychiatric disorders.

Anxiety seriously affects the quality of life negatively. The general picture that emerged in a study shows that anxiety impairs quality of life and social functionality in many areas of life. Brown and Roose found that anxiety and depression negatively affect quality of life psychologically and socially. In a study conducted by Çivi et al., when the mean quality of life scores and depression levels were compared, the mean quality of life scores of individuals with depression were found to be significantly lower than those without depression. In the study of Voelkerin and in the systematic review of Kolotkin and Andersen, it was stated that obesity reduces the quality of life. It is necessary to reduce the symptoms of depression and anxiety, to lose weight in a healthy way and to increase the quality of life.

In a study conducted by Ergen, it is recommended that respiratory exercises be routinely applied for the management of anxiety in the postoperative period. In a study by Yekta on mastectomy candidates, rhythmic breathing was found to be effective in reducing anxiety. Yusuf et al. In a study conducted by, it was determined that deep breathing exercise after surgery is an effective, inexpensive, easy and safe method in reducing the level of anxiety.

Holding the breath for a while allows the body to renew its oxygen. The 4-7-8 breathing technique provides the needed oxygen support to organs and tissues and helps to expel CO2. In the 4-7-8 breathing technique, inhale for 4 seconds, hold the breath for 7 seconds and exhale for 8 seconds. Such practices reduce anxiety by both distracting and providing relaxation by oxygenating and expelling the CO2 accumulated in the body.30 There is only one study on the 4-7-8 breathing technique. In the study of Pandekar et al., it was seen that the 4-7-8 breathing technique was effective in reducing anxiety and depression in moderate COPD patients.

It is the nurse's responsibility to provide a comfortable environment for the patient and to increase the quality of life standards. In addition, many studies show that the rate of use of non-pharmacological methods, which are the responsibility of nurses, is low. In this study, we predict that non-pharmacological deep breathing exercises and 4-7-8 breathing techniques will help reduce anxiety and increase the quality of life of patients undergoing bariatric surgery. It is the first study on the subject. This study was carried out to determine the effect of deep breathing exercise and 4-7-8 breathing technique on anxiety level and quality of life after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older - 65 years or younger
* Being on the 1st postoperative day
* Have had bariatric surgery
* No communication barrier
* Have an ASA Score I or II

Exclusion Criteria:

* Presence of major depression or psychosis
* Having a communication barrier
* Being transferred to another unit
* Leaving work voluntarily

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Inventory | Change from State and Trait Anxiety Inventory at 24 hours
  The state anxiety scale requires the person to answer at a certain moment and under certain conditions, while the trait anxiety scale requires the person to answer according to how he or she usually feels.
  This scale, which is a self-evaluation scale, consists of state anxiety and trait anxiety sections. It consists of a total of 40 questions, 20-20 in both. This scale is likert type and is graded as 'not at all-somewhat-very-completely'. The points that can be obtained from this inventory are minimum 20 and maximum 80 points.
  The scores obtained from the scale are interpreted as increasing the level of anxiety as it approaches 80, and the low level of anxiety as it approaches 20. It is interpreted in the same way when sorting by percentile.
Obese-Specific Quality of Life Scale | Change from Quality of Life at 24 hours
  This scale is a 17-item Likert-type scale scored between 0-6. According to the numerical increase order, it is expressed as 'Not at all, Hardly at all, Little, Moderate, Quite, A lot, Extremely'. The scale has no sub-dimensions. The scores obtained from all items of the scale are added together and 17 is subtracted from the obtained score. This score is divided by 102 and multiplied by 100. It is interpreted as the higher the score, the higher the quality of life, and the lower the score, the lower the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aktas GK, Ilgin VE. The Effect of Deep Breathing Exercise and 4-7-8 Breathing Techniques Applied to Patients After Bariatric Surgery on Anxiety and Quality of Life. Obes Surg. 2023 Mar;33(3):920-929. doi: 10.1007/s11695-022-06405-1. Epub 2022 Dec 8. PMID 36480101